CLINICAL TRIAL: NCT07309783
Title: Personalised EIT-guided Ventilation Strategy Versus Conventional Protective Ventilation Strategy in ARDS Patients: a Multicenter, Randomized, Controlled triaL
Brief Title: Lung EIT Image Guide Ventilation in ARDS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEARL
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
Keywords: ARDS; EIT-guided ventilation strategy; EIT-guided prone positioning; EIT-guided PEEP setting; RCT
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIT-guided group (Experimental): Prone positioning and PEEP titration guided by China-manufactured EIT.
  Interventions: Other: Recruitment maneuver and PEEP setting guided by EIT; Behavioral: Prone positioning guided by EIT
- Control group (Active Comparator): PEEP set guided by conventional PEEP-FiO₂ table and prone positioning guided by routine clinical indications without EIT guidance.
  Interventions: Other: PEEP setting according to routine practice; Behavioral: Prone positioning according to routine practice

INTERVENTIONS:
Other: Recruitment maneuver and PEEP setting guided by EIT — The EIT-guided group, will receive recruitment maneuver and PEEP titration guided by EIT to determine the optimal PEEP level.
  Arms: EIT-guided group
Other: PEEP setting according to routine practice — The control group will receive routine ventilation strategy. Routine recruitment maneuver is not recommended but may be used as rescue therapy. PEEP is set using the conventional PEEP-FiO₂ table.
  Arms: Control group
Behavioral: Prone positioning guided by EIT — The EIT-guided group, will determine prone positioning therapy based on EIT.
  Arms: EIT-guided group
Behavioral: Prone positioning according to routine practice — The control group will determine prone positioning therapy based on routine practice.
  Arms: Control group

SUMMARY:
The goal of this multi-center randomized controlled clinical trial is to learn if an individualized, bedside electrical impedance tomography (EIT)-guided ventilation strategy (including EIT-guided prone positioning and PEEP titration) can improve outcomes compared with a conventional lung-protective ventilation strategy in adult patients with acute respiratory distress syndrome (ARDS).

The main questions it aims to answer are:

Does the individualized EIT-guided ventilation strategy reduce 28-day mortality in ARDS patients? Researchers will compare the EIT-guided intervention arm to a control arm receiving routine lung-protective ventilation (without bedside EIT guidance) to see if the EIT-guided approach lowers 28-day mortality and improves other clinical outcomes.

Adult ARDS patients who meet inclusion criteria will be assigned to EIT-guided group and control group through stratified randomization:

EIT-guided group: Undergo bedside EIT assessments using a China-manufactured EIT device to guide decisions about prone positioning and individualized PEEP titration (including a recruitment maneuver).

Control group: Receive PEEP setting per conventional PEEP-FiO₂ tables and prone positioning per standard clinical indications without EIT guidance.

Both groups: Receive standard supportive ICU care and routine outcome assessments at multiple time points.

Primary outcome: 28-day mortality. Other outcomes include ventilator-free days to day 28 and so on.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ARDS receiving mechanical ventilation who meet the following diagnostic criteria:

  1. Triggered by acute risk factors such as pneumonia, non-pulmonary infection, trauma, transfusion, aspiration, or shock. Pulmonary edema is not entirely or predominantly attributable to cardiogenic causes or fluid overload, and hypoxemia/gas exchange impairment is not mainly due to atelectasis. However, ARDS can be diagnosed in the presence of these conditions if predisposing risk factors exist.
  2. Acute onset or worsening of hypoxemic respiratory failure within 1 week of the identified risk factor or onset of new or worsening respiratory symptoms.
  3. Bilateral opacities on chest radiograph or CT, or bilateral B-lines and/or consolidation on ultrasound, not fully explained by effusion, atelectasis, or nodules/masses.
  4. PaO₂/FiO₂ ≤ 300 mm Hg or SpO₂/FiO₂ ≤ 315 (if SpO₂ ≤ 97%).
* ARDS onset within 1 week.
* Mechanical ventilation ≤ 72 hours.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* Contraindications to EIT application (e.g., local skin lesions, cardiac pacemaker).
* Contraindications to prone positioning (e.g., increased intracranial pressure, intra-abdominal hypertension, spinal fractures).
* Evidence of barotrauma such as pneumothorax, mediastinal emphysema, or subcutaneous emphysema.
* End-stage disease.
* Informed consent not signed by legal guardians or family.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2028-12-20 (Estimated); Study Completion 2029-06-20 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | Day 28 after randomization
  The survival status on the 28th day after randomization

SECONDARY OUTCOMES:
Ventilator-free days within 28 days after randomization | within 28 days after randomization
  Ventilator-free days within 28 days after randomization
Ventilator-free days within 14 days after randomization | Within 14 days after randomization
  Ventilator-free days within 14 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Huaiwu He, MD, Study Chair — Department of Critical Care Medicine, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Department of Critical Care Medicine, Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China